CLINICAL TRIAL: NCT04643860
Title: A New Point-of-care Test Based on Differential Leucocyte Count, Suitable for a Mass Screening Program to Detect SARS-CoV-2: A Diagnostic Accuracy Study
Brief Title: Differential Leucocyte Count and Covid-19 Diagnosis
Status: Withdrawn | Type: Observational
Why Stopped: No patients arruoled
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: DEP_042020
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2 Infection Covid19
Keywords: SARS-CoV-2 Leucocyte General population
MeSH Terms: interventions — Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample will be taken for testing the leucocytes count to identified the presence of SARS-CoV-2 and blood drawing (3 ml) for hematological cytometric analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population: Subjects, at low and high risk of SARS-Cov-2, who undergo the nasopharyngeal swab procedure for the diagnosis of SARS-CoV-2 infection will be consecutively recruited at the Clinic Laboratory of IRCCS Neuromed in Pozzilli and Diagnostica Medica Spa in Avellino, Italy.
  Interventions: Diagnostic Test: Differential Leucocyte Count (CLDC) device and algorithm

INTERVENTIONS:
Diagnostic Test: Differential Leucocyte Count (CLDC) device and algorithm — Boold sample that detecting the early rise in leukocyte levels which has a characteristic set of ratios of leukocyte types, which identify the viral pathogen and distinguish it from a number of others. This test allows prediction of positives from full blood count results.

SUMMARY:
To date, the diagnosis of SARS-CoV-2 infection is made by identifying the viral RNA in samples collected through a nasopharyngeal swab or other respiratory samples but this technique, has several limitations for its application in a mass screening. Recently, it has been developed a new method of acquitting the occurrence of severe Sar-COV-2 infection, detecting the early rise in leukocyte levels which has a characteristic set of ratios of leukocyte types, which identify the pathogen. Primary aim of the Diagnostic Accuracy study is to validate the use of the point-of-care characteristic Differential Leucocyte Count (CLDC) device and algorithm to detect SARS-CoV-2 infection as a preliminary approach to a mass screening program. Secondary aims are to define if CLCD methods is able to detect SARS-CoV-2 infection earlier as compared to swab molecular testing.

Subjects at low and high risk of Sar-Cov-2 infection will be tested, at the same time of the nasopharyngeal swab procedure in the morning, each recruited subject will be also tested using CLDC device and algorithm. On a voluntary base, subjects will also undergo blood drawing (3 ml) for hematological cytometric analyses, research personnel will administer a questionnaire on COVID 19 symptoms and risk factors and for contact traicing. Subjects testing positive on either CLDC test but negative at the swab will undergo on a voluntary basis new swab testing after two, 5 and possibly 8 days if still negative.

It estimates to find between 150 and 200 positives in a population of 1000 subjects at different risk of infection.

DETAILED DESCRIPTION:
Introduction. In June 3rd, 2020, the Italian government started the so-called "Phase 2", which included the re-opening of working and social activities. In this framework, the issue of how to identify the asymptomatic individuals who, unwittingly, can spread SARS-CoV-2 infection and pose a threat to public health has been raised worldwide. The mondial population are now experiencing the phase 3 of the pandemic with a rapid increase in the spreading of infection and in the occurrence of new cases. It is now imperative to guarantee the health and safety of the people called back to work and to create a safety protocol in commercial and meeting spaces, which means preventing infected people from causing new epidemic outbreaks. For this purpose, a well-established mass screening program is required to meet several needs: first, it should provide the result in a few minutes, it should be easily delivered on the territory, non-medical healthcare professionals should perform it in a simple way also, and should be non-invasive, repeatable and reliable.

To date, the diagnosis of SARS-CoV-2 infection is made by identifying the viral RNA in samples collected through a nasopharyngeal swab or other respiratory samples. This technique, however, has several limitations for its application in a mass screening, among which the most important ones are the time necessary for the diagnosis, the crowding of those centers appointed to analyze the specimens, and the non-negligible risk of viral transmission to the healthcare workers.

Point-of-care testing with rapid turnaround times would allow more effective triage in settings where patient management and infection control decisions need to be made rapidly.

Recently, it has been developed a new method of acquitting the occurrence of severe Sar-COV-2 infection and resulting COVID-19, detecting the early rise in leukocyte levels which has a characteristic set of ratios of leukocyte types, which identify the viral pathogen and distinguish it from a number of others. This test allows prediction of positives from full blood count results, sensitive up to 14 days earlier than real-time quantitative PCR (RT-qPCR), at a cost at least an order of magnitude lower than other tests such as RT-qPCR and antibody tests.

Aim of the study. Primary aim of the Diagnostic Accuracy study is to validate the use of the point-of-care characteristic Differential Leucocyte Count (CLDC) device and algorithm to detect SARS-CoV-2 infection in both symptomatic and asymptomatic individuals as a preliminary approach to a mass screening program. The comparison is represented by the nasopharyngeal swab molecular testing, the gold standard of COVID-19 diagnosis, for algorithm validation and hematological cytometric analyses by Coulter HMX, Beckman Coulter, for device validation.

Secondary aims are to define if CLCD methods is able to detect SARS-CoV-2 infection earlier as compared to swab molecular testing and to perform a contact tracing study on all double-positive patients to estimate their original date of infection to determine the curve of test sensitivity against initial infection.

Methods. Subjects who undergo the nasopharyngeal swab procedure for the diagnosis of SARS-CoV-2 infection will be consecutively recruited at the Clinic Laboratory of IRCCS Neuromed in Pozzilli and Diagnostica Medica Spa in Avellino, Italy. Subjects at low and high risk of Sar-Cov-2 infection will be tested: healthcare workers, patients to be electively hospitalization for reason other than COVID-19 or other infectious disease, persons who had direct contact with infected patients.

At the same time of the nasopharyngeal swab procedure in the morning, each recruited subject will be also tested using CLDC device and algorithm (CLCD 2). On a voluntary base, subjects will also undergo blood drawing (3 ml) for hematological cytometric analyses by Coulter HMX, Beckman Coulter and will be tested using only CLDC algorithm (CLCD 1).

The outcome assessors are blinded, since the results of the rRT-PCR analysis require at least 6 hours before being available. Research personnel will administer a questionnaire on COVID 19 symptoms and risk factors and for contact traicing (day, mode) Subjects testing positive on either CLDC test but negative at the swab will undergo on a voluntary basis new swab testing after two, 5 and possibly 8 days if still negative.

Independent blinded clinicians through real-time reverse transcription (rRT)-PCR, will analyse the nasopharyngeal swab accordingly to the International guidelines.

For device validation, Full Blood Count (FBC) will be analyzed both by measuring Full Blood Count and entering the results into the Medichain CLDC-1 portal for rapid analysis and through the point-of-care device connected to the smart-phone (the Medichain CLDC-2 smartphone microscope - the Adstock Test).

The Medichain CLDC-2 smartphone microscope, a device that clip onto a standard smartphone will be used to analyse drops of blood of approximately 1µl smeared on a microscope slide (version 2 - Adstock Test) illuminated in phase-contrast mode. Images will then be sent from the devices to Medichain for analysis on servers in the UK and manual cross-checking.

Then a preparatory algorithm Athena S3ER capable of measuring input specific FBC parameters analyzes data from this result and returning an output; taking into account abnormal occurrence in numbers of specific FBC parameters at the onset of infection. The basic test portal for this study (known as the S3ER algorithm) would be at http://cldc.medichain.online. The preferred extended portal is the research portal at http://cldc.medichain.online/research Nasopharyngeal swab analysis. Samples will be subjected to viral thermal inactivation for 1 minute at 90 °C. RNA extraction from the nasopharyngeal swab will be performed with the Abbott mSample Preparation System (Promega corporation) and an automated extraction system (Extraction m2000SP, Abbott Molecular). The extracted RNA will be amplified with GeneFinderTM COVID19 Plus RealAmp PCR kit (ELITechGroup), a one-step rRT-PCR system targeting SARS-CoV-2 RdRp, E, and N genes. All recruited subjects will undergo the nasopharyngeal swab, thus Partial verification bias will beabsent. The CLDC test and nasopharyngeal swab procedures will be performed at the same moment to avoid disease progression bias. Being the CLCD test and the nasopharyngeal swab analyzed by independent blinded clinicians, information bias will be avoided when interpreting the rate-PCR results of the swabs. The index test is completely independent of the reference test, so to avoid the Incorporation bias. Inconclusive results will be recorded.

Sample size and statistical analysis. The incidence of positivity for COVID-19 is presently estimated at 15% in the general population and 20% in high-risk people. Therefore, it estimates to find between 150 and 200 positives in a population of 1000 subjects at different risk of infection.

A sample size of 1000 with a prevalence of 15% of positive nasopharyngeal swabs would suffice to estimate a sensitivity of around 0.75 with a precision of 0.15 for the 95% confidence interval and a power of 0.8.

Demographic and clinical features of the eligible participants will be summarized by using mean and standard proportion, or absolute and relative frequencies, for continuous and discrete variables, respectively. For descriptive purposes only, the same statistical analyses will be reported also in positive and negative nasopharyngeal swab subjects. In case of technical failure of testing without the possibility to repeat the procedure, the participants will be excluded from further analyses. In the other subjects, the sensitivity and specificity for the CLDC (index test) when compared to the nasopharyngeal swab (reference test 1) or to FBC (reference test 2) will be estimated, and their 95% confidence interval will be calculated from the exact binomial distribution. These analyses will be also replicated according to main subject characteristics. The participants will be characterizing as true positives (TP), false positives (FP), as well as false negatives (FN) and true negatives (TN), in terms of prevalence of positive CLDC-PCR, CLDC-FBC results. The null association of no difference across TP, FP, FN and TN will test using a Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Signing a written consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects at low and high risk of Sar-Cov-2 infection, who undergo the nasopharyngeal swab procedure for the diagnosis of SARS-CoV-2 infection will be consecutively recruited at the Clinic Laboratory of IRCCS Neuromed in Pozzilli and Diagnostica Medica Spa in Avellino, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
validation | 4 months
  Primary aim is to validate the use of the point-of-care characteristic Differential Leucocyte Count (CLDC) device and algorithm to detect SARS-CoV-2 infection as a preliminary approach to a mass screening program.

SECONDARY OUTCOMES:
test sensitivity | 4 months
  Secondary aims are to define if CLCD methods is able to detect SARS-CoV-2 infection earlier as compared to swab molecular testing and to perform a contact tracing study on all double-positive patients to estimate their original date of infection to determine the curve of test sensitivity against initial infection.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS, Italy